CLINICAL TRIAL: NCT05324397
Title: Safety and Efficacy Study of the Neurent Medical NEUROMARK™ System in Subjects With Chronic Rhinitis - A Prospective, Single-arm, Multicenter Clinical Study
Brief Title: Safety and Efficacy Study of the Neurent Medical NEUROMARK™ System in Subjects With Chronic Rhinitis (CLARITY)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Neurent Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIP-0006
Record Dates: First submitted 2022-04-04; First posted 2022-04-12 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Chronic Rhinitis
Keywords: Rhinitis
MeSH Terms: conditions — Rhinitis

STUDY DESIGN:
Intervention Model Description: A prospective, single-arm, multicenter clinical study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Experimental: Treatment (Experimental): Subjects will undergo treatment with the NEUROMARK System
  Interventions: Device: NEUROMARK System

INTERVENTIONS:
Device: NEUROMARK System — The NEUROMARK™ System is indicated for use in otorhinolaryngology (ENT) surgery for creation of radiofrequency (RF) lesions to disrupt posterior nasal nerves in patients with chronic rhinitis.

SUMMARY:
The CLARITY Study is a prospective, single-arm, multicenter safety and efficacy study of the Neurent Medical NEUROMARK System in subjects with chronic rhinitis.

ELIGIBILITY:
Inclusion Criteria:

* Subject provides written informed consent, including authorization to release health information.
* Subject is 18 years of age or older at the time of consent.
* Subject has provided a negative pregnancy test (if subject is a woman of childbearing potential (WOCBP).
* Subject WOCBP must be practicing and willing to continue an effective method of birth control during the course of the study.
* Confirmation of moderate to severe symptoms of rhinorrhea. (VAS NSS score for runny nose ≥ 5.0 and rTNSS score for runny nose ≥ 2).
* Confirmation of mild to severe symptoms of nasal congestion. (VAS NSS score ≥ 2.5 for stuffy nose (congestion) and rTNSS score of ≥ 1).
* Confirmation that the total combined VAS NSS score is ≥ 10 for nasal congestion and runny nose.
* Subjects stated willingness to comply with all study procedures, post- treatment care and availability for the duration of the study follow up of 1 year.
* Subject tests negative for active COVID-19 at the start of study screening and continues to be free from COVID-19 symptoms until the time of enrollment/treatment.
* Subject understands and agrees to follow local COVID-19 restrictions (social distancing, face mask, etc.).
* Nasal anatomy appropriate to receive the NEUROMARK™ System.
* Subject is experiencing long term chronic rhinitis. Subject has been experiencing symptoms of rhinitis for at least 6 months prior to enrollment, defined as: rhinorrhea, anterior runny nose AND congestion, blockage (stuffy nose, obstruction).

Exclusion Criteria:

* Subject has clinically significant anatomic obstruction that limits access to the posterior nose as determined by the Study Investigator such as severe septal deviation, prior surgical considerations, cleft palate, nasal polyps, or sino-nasal tumor.
* Subject has an active nasal or sinus infection at the time of treatment.
* Subject has a diagnosis of Atrophic Rhinitis.
* Subject has a Lund-Mackay score >3 during the screening phase, an active history of chronic sinusitis (within the last year).
* Subject has a septal perforation or nasal mucosal erosion/ulceration.
* Subject experiences numbness of the soft palate, excessive dry eye, excessive dry nose, or other indication of neuro/nerve compromise in the sino-nasal anatomy.
* Subject has had prior sinus or nasal surgery that may prevent access or proper placement of the NEUROMARK™ System.
* Subject has had prior head or neck irradiation (head/neck cancer therapy).
* Subject has an allergy or intolerance to anaesthetic agent or other study-required materials.
* Subject is taking anticoagulant medication or 325 mg aspirin that cannot be discontinued before the procedure and for the length of the study.
* Subject has a history of nasal manifestation of rheumatic disease.
* Subject has started a new sino-nasal medication regimen within 4 weeks prior to treatment (i.e. antihistamines, cromolyn, leukotriene receptor antagonists, inhaled or systemic steroids, anticholinergics, expectorants, decongestants) that, per the manufacturer's labelling, has not yet stabilized.
* Subject has uncontrolled Hypothyroidism.
* Subject has uncontrolled Hypertension (stage 2 or higher).
* Subject is an active smoker or has been a smoker within the last 6 months (patient reported).
* Any physical condition that in the Investigator's opinion would prevent adequate study participation or pose increased risk to the study Subject.
* Subject is pregnant, nursing or plans to become pregnant during the study, or is a WOCBP, but is not willing to use an effective method of birth control.
* Patient is enrolled in an investigational drug or device study or has participated in such a study within the last 30 days prior to screening that in the opinion of the Investigator would interfere with the study results.
* Patient presents with any condition or situation which, in the Investigator's opinion, puts the Subject at risk, could confound the study results, or may interfere significantly with the Subject's participation in the study.
* Subject presents with acute sinusitis at time of treatment or other sino-nasal related illness other than rhinitis.
* Subject has history of chronic epistaxis or nosebleed episodes within the last 12 months.
* Subject has rhinitis symptoms due to seasonal allergies only.
* Subject has received previous procedure or surgery for chronic rhinitis and/or to disrupt the posterior nasal nerve.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2022-03-14 (Actual); Primary Completion 2023-10-04 (Actual); Study Completion 2023-10-04 (Actual)

PRIMARY OUTCOMES:
Safety | 1 month
  Safety will be evaluated based on frequency of Serious Adverse Events (SAEs) directly attributable to the NEUROMARK System at one (1) month post index procedure.
Efficacy | 3 months
  Efficacy will be assessed by the change in Visual Analog Scale (VAS) Nasal Symptom Score (NSS) from baseline through 3 months for rhinorrhea and nasal congestion

CONTACTS AND LOCATIONS:
Overall Officials: Annalise Sorensen, Study Director — Neurent Medical
Locations (4):
- United States (4):
  - Alabama Nasal and Sinus Center, Birmingham, Alabama
  - Centers for Advanced ENT Care, Baltimore, Maryland
  - Specialty Physician Associates, Bethlehem, Pennsylvania
  - ENT & Allergy Associcates, Puyallup, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Reh DD, Lay K, Davis G, Dubin MG, Yen DM, O'Malley EM, Sillers M. Long-term outcomes following impedance-controlled radiofrequency ablation for the treatment of chronic rhinitis. Laryngoscope Investig Otolaryngol. 2024 Jun 4;9(3):e1286. doi: 10.1002/lio2.1286. eCollection 2024 Jun. PMID 38835333
- [Derived] Reh DD, Lay K, Davis G, Dubin MG, Yen DM, O'Malley EM, Sillers M. Clinical evaluation of a novel multipoint radiofrequency ablation device to treat chronic rhinitis. Laryngoscope Investig Otolaryngol. 2023 Mar 16;8(2):367-372. doi: 10.1002/lio2.1040. eCollection 2023 Apr. PMID 37090860